CLINICAL TRIAL: NCT06323213
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of 610 in Chinese Adult Subjects With Severe Eosinophilic Asthma
Brief Title: Efficacy and Safety Study of 610 in Patients With Severe Asthma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSGJ-610-BA-III-01
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 610 group (Experimental): Subjects will receive 610 for 52 weeks.
  Interventions: Drug: 610
- placebo group (Placebo Comparator): Subjects will receive placebo for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 610 — 610 subcutaneously injection.
  Arms: 610 group
Drug: Placebo — Placebo subcutaneously injection.
  Arms: placebo group

SUMMARY:
The primary objective of the study is to evaluate the efficacy and safety of 610 in Chinese adults with severe asthma.

DETAILED DESCRIPTION:
The total duration of study per patient is approximately 66 weeks, including 6 weeks of screening period, 52 weeks of treatment period and 8 weeks of follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent prior to participation in the study.
2. Male or female adults ages 18 to 75 years old when signing the informed consent.
3. Documented diagnosis of asthma for at least one year prior to screening.
4. History of physician-diagnosed asthma requiring treatment with ICS and at least one other control medication for at least 6 months prior to screening.

Exclusion Criteria:

1. Presence of a known pre-existing, clinically important lung condition other than asthma.
2. Severe asthma exacerbation within 4 weeks prior to randomization.
3. Subjects with any eosinophilic diseases other than asthma.
4. Known, pre-existing severe or clinically significant cardiovascular disease.
5. known, pre-existing other concurrent clinically significant medical conditions that are uncontrolled with standard treatment.
6. Subjects who have active Hepatitis B, Hepatitis C or HIV infections as determined by positive results at Screening.
7. Subjects with allergy/intolerance to a monoclonal antibody.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of severe exacerbation events | Up to 52 weeks
  Annualized rate of severe exacerbation events during the 52-week placebo-controlled treatment period

SECONDARY OUTCOMES:
Time to first severe exacerbation event | Up to 52 weeks
  Time to first severe exacerbation event during the 52-week placebo-controlled treatment period
Annualized rate of severe exacerbation events resulting in hospitalization or emergency room visit | Up to 52 weeks
  Annualized rate of severe exacerbation events resulting in hospitalization or emergency room visit during the 52-week placebo-controlled treatment period
Change from baseline in ACQ score | Up to 52 weeks
  Change from baseline to week 52 in ACQ score
Change from baseline in ST. GEORGE'S Respiratory Questionnaire(SGRQ) | Up to 52 weeks
  Change from baseline to week 52 in SGRQ score
Change in pre-bronchodilator forced expiratory volume (FEV1) | Up to 52 weeks
  Absolute change from baseline to week 52 in pre-bronchodilator FEV1
Assessment of adverse events (AEs) | Up to 60 weeks
  Number of participants with adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhang, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Xin Zhou, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China